CLINICAL TRIAL: NCT02723565
Title: Ultrasound to Evaluate Failure of Liberation From Mechanical Ventilation
Acronym: USEFUL
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ewan Goligher, Intensivist, University Health Network, Toronto
Other Study IDs: 14-7400-B
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Acute Respiratory Failure; Respiration, Artificial; Weaning
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the heart, lungs and diaphragm of patients who fail a trial of spontaneous breathing to determine the physiological mechanism of weaning failure.

DETAILED DESCRIPTION:
The transition to unassisted breathing after invasive ventilation often proves challenging, with over 40% of patients failing their first attempt of unassisted breathing. Persistent ventilator dependence predisposes patients to nosocomial complications and increases the economic burden of critical illness. Ventilator-dependence results from an imbalance between the load and capacity of the respiratory muscle pump. Patients who fail a trial of spontaneous breathing commonly exhibit excess respiratory loads secondary to weaning-induced pulmonary edema, atelectasis or dynamic hyperinflation. Many patients who are dependent on the ventilator also show a striking loss of pump capacity due to diaphragm dysfunction. Though each of these mechanisms respond to specific interventions, it is often difficult for physicians to discern which mechanisms are at play at the bedside. Bedside ultrasound is a potentially useful means of evaluating cardiac, pulmonary and diaphragm function during weaning failure. It is readily available, highly feasible and already widely employed in clinical practice. As yet, no study has evaluated the accuracy and feasibility of combining echocardiography with lung and diaphragm ultrasound to comprehensively evaluate the physiological mechanisms of weaning failure. The objectives of this study are to establish the utility of a rapid thoracic ultrasound exam to diagnose mechanisms of ventilation liberation failure and to assess the relationship between cardiothoracic variability during spontaneous breathing and different physiological mechanism of weaning failure.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age receiving invasive mechanical ventilation for at least 24 hours
* patients who fulfill standard criteria for readiness for a trial of spontaneous breathing (no or minimal sedation, patient awake and interactive; minimal vasopressor/inotrope requirements (Norepinephrine < or = 0.1, Dopamine < 10, Vasopressin/Epinephrine off); fraction of inspired oxygen < or = 50%; spontaneous inspiratory efforts as indicated by patient-triggered breaths; positive end-expiratory pressure < or = 10 cm H20)
* patients who fail a trial of spontaneous breathing (transient reduction of ventilator support for any duration up to 2 hours as per local ICU practice - typically PS 5 with PEEP 5 OR CPAP 5 OR T-piece)

Exclusion Criteria:

* patients with a coagulopathy (INR > 2.5, platelet count < 30x10^6/L) or previously diagnosed bleeding diathesis or are receiving anticoagulant drugs at therapeutic doses (ie. excluding venous thromboembolic prophylaxis)
* patients with a contraindication to nasogastric tube insertion (esophageal varices, upper GI tract surgery, facial trauma, etc.)
* patients receiving extra-corporeal life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity for diagnosis of physiological mechanisms causing weaning failure | Physiological measurements for diagnostic classification measured simultaneously with ultrasound measurements
  Mechanisms responsible for weaning failure will be diagnosed by field experts using clinical data collected from the chart along with physiological measurements (respiratory mechanics, maximal inspiratory pressure, markers of pulmonary edema including changes in serum total protein and BNP and central venous pressure). The diagnosis derived from a pre-specified ultrasound-based classification system will be compared to the gold standard expert-derived diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan C Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No